CLINICAL TRIAL: NCT00753519
Title: Intermittent Theta-Burst Transcranial Magnetic Stimulation (TBS) for the Treatment of Parkinson Disease
Brief Title: Transcranial Magnetic Stimulation to Treat Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mark Hallett (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Mark Hallett, Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080212; 08-N-0212
Record Dates: First submitted 2008-09-13; First posted 2008-09-16 (Estimated); Results first posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Brain Stimulation; Motor Cortex; Bradykinesia; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease; Hypokinesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real iTBS (Experimental): iTBS is a novel form of excitatory rTMS that may induce larger and longer lasting changes that standard rTMS. iTBS consists of bursts of 3 pulses at 50 Hz repeated at 200 msec intervals. The 2 sec trains were repeated 20 times every 10 sec. iTBS was applied to the primary motor and the dorsolateral prefrontal cortex bilaterally.
  Interventions: Device: Real iTBS
- Sham iTBS (Sham Comparator): The sham coil was placed in the same areas, and made a similar sound as the rTMS but was without a magnetic pulse.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: Real iTBS — Real iTBS was performed in 8 sessions over 2 successive weeks, a session/day for 4 consecutive days/week.
  Arms: Real iTBS
Device: Sham iTBS — Sham iTBS was performed in 8 sessions over 2 successive weeks, a session/day for 4 consecutive days/week.
  Arms: Sham iTBS

SUMMARY:
This study will look at the effects of transcranial magnetic stimulation (TMS) on symptoms of Parkinson's disease. TMS is a method of brain stimulation that may be able to change the activity of the nerve cells of the brain. This study will examine the effects of a specific pattern of stimulation called intermittent theta-burst TMS (iTBS), which uses repeated magnetic pulses delivered in short bursts.

People with mild to moderately severe Parkinson's disease who are between 40 and 80 years of age and whose main problems are slow movement and stiffness may be eligible for this study.

Participants undergo the following tests and procedures:

* Random assignment to real or placebo (sham) iTBS treatment.
* iTBS sessions (real or sham) 4 times a week for 2 consecutive weeks. For this test, the subject sits in a comfortable chair. A wire coil is held on the subject's scalp, and a brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in the muscles of the face, arm or leg.
* Test of gait (walk), hand and arm movements before and after each session. The gait test requires walking 10 meters (about 30 yards) in the same corridor with the same shoes.
* Extended testing. The first and last gait tests (done before starting iTBS and after the eighth session) require coming off any Parkinson's medication for at least 12 hours before the test. On these test days, subjects also undergo a clinical examination, short neuropsychological test battery, a computer-based reaction time test and depression and quality-of-life rating scales. These procedures are repeated in a follow-up visit 1 month after the last session.

DETAILED DESCRIPTION:
Objective

To demonstrate cumulative and long-lasting improvement of parkinsonian symptoms by iTBS and its safety in PD patients.

Study population

Patients (40-80 years of age) with PD, Hoehn and Yahr disease stage of 2 to 4 while off, being on a regimen including levodopa with a total dose of medication equal to more than 300 mg of levodopa, including their dopamine agonist agents, and having problems with walking and needing 6 seconds or more to walk a 10-meter distance.

Design

Randomized, double-blind, placebo (sham)-controlled study. Enrollment of 30 patients with PD in 2 groups (real versus sham stimulation). Performance (8 interventions) of iTBS with large circular coil over motor and prefrontal cortex on both sides. Assessment with standard tests of motor function over a one-month period.

Outcome measure

The primary endpoint is change in gait speed as assessed by the time it takes to walk 10 m.

Secondary endpoints include changes in bradykinesia as assessed by measuring the time it takes to do ten combined hand and arm movements, and in total and motor UPDRS score.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Men and women aged 40 to 80 years with DOPA-responsive PD
* Hoehn and Yahr grade of 2 to 4 while off
* Must be on a regimen including levodopa.
* Total dose of levodopa and dopamine agonists (using dopamine equivalents) has to be equal to or more than 300 milligrams per day
* Problems with walking, including freezing gait time for a 10-meter distance greater than six seconds or more

EXCLUSION CRITERIA:

* Any active psychiatric disease or evidence of dementia
* History of seizures and epilepsy
* Concurrent use of tricyclic antidepressants, neuroleptic agents, or any other licit or illicit drugs other than anti-parkinsonian agents that could lower the seizure threshold except for SSRI
* Pallidotomy, implanted electrodes and generator for deep brain stimulation
* Pregnancy
* Surgically or traumatically implanted foreign bodies such as a pacemaker, implanted medical pump, implanted hearing aids, metal plate in the skull, or metal implant in the skull or eyes (other than dental appliances or fillings) that may pose a physical hazard during TEP.
* Study would cause undue risk or stress for reasons such as tendency to fall, excessive fatigue, general frailty, or excessive apprehensiveness.
* Dementia as assessed by the Folstein's Mini-Mental Test Examination (MMSE less than or equal to 24/30) or mentally impaired patients having no capacity to provide their own consent (the physician establishing the diagnosis and applying UPDRS will evaluate patient's mental capacity using conventional clinical interview)
* Unable to walk a 10-meter distance.
* More than occasional falls, i.e. daily falls (corresponding to a score greater than or equal to 3 and more in UPDRS item 13), history of fall(s) with significant injuries, absence of postural response in the on condition and/or spontaneous loss of balance in the off condition (corresponding to a score of greater than or equal to 2 and greater than or equal to 3 in on/off condition, respectively, in UPDRS item 30)

Pregnancy is unusual in patients with PD, grade 2-4. Urine sample for the pregnancy test will be obtained in patients of childbearing potential prior to the iTBS start, at the day of the initial interview and signing the consent form. Women of childbearing potential will be asked to take appropriate measures to prevent a pregnancy during the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aarsland D, Larsen JP, Waage O, Langeveld JH. Maintenance electroconvulsive therapy for Parkinson's disease. Convuls Ther. 1997 Dec;13(4):274-7. PMID 9437571
- [Background] Baudewig J, Siebner HR, Bestmann S, Tergau F, Tings T, Paulus W, Frahm J. Functional MRI of cortical activations induced by transcranial magnetic stimulation (TMS). Neuroreport. 2001 Nov 16;12(16):3543-8. doi: 10.1097/00001756-200111160-00034. PMID 11733708
- [Background] Belmaker RH, Grisaru N. Magnetic stimulation of the brain in animal depression models responsive to ECS. J ECT. 1998 Sep;14(3):194-205. PMID 9773358

RESULTS

PARTICIPANT FLOW:
Groups:
- Real iTBS: iTBS is a novel form of excitatory rTMS that may induce larger and longer lasting changes than standard rTMS. iTBS consists of bursts of 3 pulses at 50 Hz repeated at 200 msec intervals.
- Sham iTBS: Sham iTBS
Period: Overall Study
Arm/Group | Real iTBS | Sham iTBS
Started | 13 | 15
Completed | 13 | 13
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real iTBS | Sham iTBS | Total
Number analyzed (Participants) | 13 | 13 | 26
Age Continuous [Mean (Standard Deviation); unit: years] | 62.1 (6.9) | 65.6 (9.0) | 63.85 (8.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 7 | 11 | 18
Duration of disease [Mean (Standard Deviation); unit: years] | 10.8 (7.1) | 6.5 (3.4) | 8.62 (5.87)
Hoehn-Yahr "on" [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr scale is a system used to describe how the symptoms of Parkinson's disease progress. The scale ranges from 1-5 with 1 representing unilateral involvement with minimal or no functional disability and 5 representing confinement to bed or wheelchair unless aided. The Hoehn and Yahr measurement was taken while the subject was on dopaminergic medication.
  units on a scale | 2.6 (0.2) | 2.5 (0.1) | 2.52 (0.17)
Hoehn-Yahr "off" [Mean (Standard Deviation); unit: units on a scale] — The Hoehn and Yahr scale is a system used to describe how the symptoms of Parkinson's disease progress. The scale ranges from 1-5 with 1 representing unilateral involvement with minimal or no functional disability and 5 representing confinement to bed or wheelchair unless aided. The Hoehn and Yahr measurement was taken while the subject was off dopaminergic medication for 12 hours or more (overnight).
  units on a scale | 3.0 (0.4) | 2.9 (0.2) | 2.90 (0.32)
Total LED [Mean (Standard Deviation); unit: milligrams] — Total levodopa equivalent dose
  milligrams | 1180.9 (662.4) | 732.3 (344.8) | 956.6 (565.7)
Tremor [Number; unit: participants]
  Presence of tremor | 10 | 9 | 19
  Absence of tremor | 3 | 4 | 7
Gait freezing [Number; unit: participants]
  Presence of gait freezing | 10 | 3 | 13
  Absence of gait freezing | 3 | 10 | 13
Fluctuations [Number; unit: participants]
  Presence of fluctuations | 11 | 4 | 15
  Absence of flucuations | 2 | 9 | 11
Dyskinesias [Number; unit: participants] — Presence or absence of dyskinesias (diminished voluntary movements and the presence of involuntary movements).
  participants
    Presence of dyskinesias | 9 | 2 | 11
    Absence of dyskinesias | 4 | 11 | 15
Falls [Number; unit: participants]
  Presence of falls | 1 | 0 | 1
  Absence of falls | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed
Description: Gait speed was assessed by measuring the time it takes to walk 10 meters. Subject's gait speed was measured while on medication and off medication for each group, i.e., real iTBS and sham iTBS. Two trials were averaged for each condition. Patients were instructed to walk fast without taking the risk of falling, wearing the same shoes and consistently using assistive devices if needed. Gait speed was measured at baseline, 1 day post intervention, and 1 month post intervention.
Time Frame: baseline, 1 day post iTBS
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- On Medication Real iTBS: Subjects ON medication while receiving REAL iTBS
- On Medication Sham iTBS: Subjects ON medication while receiving SHAM iTBS
- Off Medication Real iTBS: Subjects OFF medication while receiving REAL iTBS
- Off Medication Sham iTBS: Subjects OFF medication while receiving SHAM iTBS
Arm/Group | On Medication Real iTBS | On Medication Sham iTBS | Off Medication Real iTBS | Off Medication Sham iTBS
Number analyzed (Participants) | 13 | 13 | 13 | 13
seconds
  baseline | 8.35 (1.98) | 8.41 (1.98) | 25.84 (26.1) | 8.80 (25.0)
  1 day post | 7.68 (2.02) | 7.96 (2.02) | 10.88 (3.81) | 8.20 (3.66)

2. Secondary Outcome: Bradykinesia
Description: Bradykinesia refers to the slowness in executing a movement. Bradykinesia was assessed by measuring the time in seconds it takes to do the following sequence, 10 times: 1) hand closing and opening while squeezing a ball 2) elbow flexion 3) hand closing and opening, and 4) elbow extension. Subjects were allowed to practice these hand and arm movements until performance appeared not to get faster, and then were abstained from further practice to minimize learning effects. The time it takes subjects to execute the entire sequence 10 times with either the left or right arm/hand was measured. Means are reported for each group.
Time Frame: baseline, 1 day post iTBS
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | On Medication Real iTBS | On Medication Sham iTBS | Off Medication Real iTBS | Off Medication Sham iTBS
Number analyzed (Participants) | 13 | 13 | 13 | 13
seconds
  baseline | 13.69 (5.33) | 13.25 (5.33) | 17.23 (8.10) | 14.20 (7.78)
  1 day post | 10.32 (3.48) | 10.88 (3.48) | 14.20 (7.78) | 10.80 (4.03)

3. Secondary Outcome: Total UPDRS Score
Description: The Total Unified Parkinson's Disease Rating Scale (UPDRS) is an overall assessment scale that quantifies the signs and symptoms of Parkinson's disease. The total UPDRS score consists of mentation, behavior, mood, activities of daily living and motor components, and ranges from 0 (not affected) to 176 (most severely affected). The total UPDRS score is obtained from patient examination, interview and patient questionnaires.
Time Frame: baseline, 1 day post iTBS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Medication Real iTBS | On Medication Sham iTBS | Off Medication Real iTBS | Off Medication Sham iTBS
Number analyzed (Participants) | 13 | 13 | 13 | 13
units on a scale
  baseline | 55.54 (15.81) | 57.15 (15.81) | 77.85 (17.05) | 65.92 (17.05)
  1 day post | 51.08 (16.37) | 47.62 (16.37) | 70.85 (16.26) | 70.85 (16.26)

4. Secondary Outcome: Motor UPDRS
Description: The Motor Unified Parkinson's Disease Rating Scale (UPDRS) includes only the motor assessment of the UPDRS (Part III) and examines speech, facial expression, tremor at rest, action tremor, rigidity, finger taps, hand movements, hand pronation and supination, leg agility, arising from chair, posture, gait, postural stability and body bradykinesia. The scores range from 0 (no motor impairment) to 108 (severe motor impairment).
Time Frame: baseline, 1 day post iTBS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | On Medication Real iTBS | On Medication Sham iTBS | Off Medication Real iTBS | Off Medication Sham iTBS
Number analyzed (Participants) | 13 | 13 | 13 | 13
units on a scale
  baseline | 32.00 (12.86) | 37.54 (12.86) | 49.00 (12.88) | 45.69 (12.38)
  1 day post | 29.08 (12.13) | 32.31 (12.13) | 43.92 (12.59) | 41.31 (12.10)

ADVERSE EVENTS:
Arm/Group | Real iTBS | Sham iTBS
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/13
Other Adverse Events (participants affected / at risk) | 1/13 | 1/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real iTBS (N=13) | Sham iTBS (N=13)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) — Myocardial infarction considered unrelated to the study
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Real iTBS (N=13) | Sham iTBS (N=13)
Transient non pulsating tinnitus (L) (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Epileptiform discharges (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No